CLINICAL TRIAL: NCT02113111
Title: The Effects of Therapeutic Fasting on Self Efficacy Measures - a Prospective Observational Trial
Brief Title: Effects of Fasting on Self Efficacy
Acronym: TheraFast
Status: Completed | Type: Observational
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Romy Lauche, Principal Investigator, Universität Duisburg-Essen
Other Study IDs: 13-5522 TheraFast
Record Dates: First submitted 2014-04-10; First posted 2014-04-14 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Pain; Fibromyalgia; Rheumatoid Arthritis; Gout; Headache; Arthritis; Gastrointestinal Diseases; Irritable Bowel Syndrome; Inflammatory Bowel Disease; Cardiovascular Diseases
MeSH Terms: conditions — Chronic Pain; Fibromyalgia; Arthritis, Rheumatoid; Gout; Headache; Arthritis; Gastrointestinal Diseases; Irritable Bowel Syndrome; Inflammatory Bowel Diseases; Cardiovascular Diseases | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fasting: Patients being admitted to an internal integrative medicine hospital and referred to therapeutic fasting therapy
  Interventions: Behavioral: Fasting

INTERVENTIONS:
Behavioral: Fasting — Fasting therapy was adapted from Buchinger, including a fasting period of 7 days. After 2 prefasting days with 800kcal per day from vegetables and rice/potatoes, fasting starts with the ingestion of an oral laxative. During fasting patients receive small quantities of juice and herbal teas, and a vegetable broth for lunch, altogether no more than 350kcal per day. At the end, fasting is broken by an apple or cooked potato, and for the following 3 days nutrition returns to normocaloric diet.

SUMMARY:
The study aims to investigate

* if a 7 day therapeutic fasting regimen will affect self-efficacy of patients with chronic diseases
* the effects of fasting on physical and mental well-being, quality of life and body awareness/image
* the association between patients characteristics and the perceived health benefit after fasting
* the association between Diagnosis according to traditional Chinese medicine and physical and mental well-being during the course of fasting
* experiences and perceptions of patients during fasting therapy

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* eligible for fasting, i.e. normal weight (no anorexia, no nutritional deficiency, no BMI<18 or >35, no eating disorder)

Exclusion Criteria:

* psychiatric disorder
* type 1 diabetes
* hepatitis
* severe somatic disorder (oncological disease, hepatological or nephrological)
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being treated in an integrative clinic for internal medicine Patients recommended for fasting therapy during the inpatient treatment
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2014-04; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Self efficacy questionnaire | up to 6 months
  Self efficacy questionnaire (SWE) by Schwarzer and Jerusalem, 1999
Bodily self-efficacy | up to 6 months
  Bodily self-efficacy (Schützler and Witt, 2013)

SECONDARY OUTCOMES:
Ability and will to change | 2 weeks, 6 months
  Ability and will to change (Büssing, 2008)
Easiness of life | 2 weeks, 6 months
  Questionnaire on emotional and physical reactions
Health-related quality of life | 2 weeks, 6 months
  Short Form (36) Health Survey
Body responsiveness | 2 weeks, 6 months
  Body Responsiveness Scale (BRS)(Daubenmier 2005)
Body awareness and dissociation | 2 weeks, 6 months
  Scale of Body Connection (SBC) (Price and Thompson 2007)
Body Awareness | 2 weeks, 6 months
  Body Awareness Questionnaire (BAQ) (Shields 1989)
Symptoms | 2 weeks, 6 months
  MYMOP questionnaire (Paterson)
Depression | 2 weeks, 6 months
  Becks Depression Inventory (BDI)
Safety | 2 weeks
  Any adverse effect during the study period

OTHER OUTCOMES:
Well-being | 2 weeks
  Daily log, visual analogue scales (VAS) on positive or negative physical or psychological states, side effects, daily rating
Diagnosis according to traditional Chinese medicine | day 1
  Assessment of traditional Chinese medicine type will be used for correlational analysis
Experiences | 2 weeks
  gathered by qualitative interviews

CONTACTS AND LOCATIONS:
Overall Officials: Gustav Dobos, Prof, Study Director — Department of Internal and Integrative Medicine, Kliniken Essen-Mitte, Faculty of Medicine, University of Duisburg-Essen; Romy Lauche, PhD, Principal Investigator — Department of Internal and Integrative Medicine, Kliniken Essen-Mitte, Faculty of Medicine, University of Duisburg-Essen
Locations (1):
- Department of Internal and Integrative Medicine, Kliniken Essen-Mitte, Essen, Germany

REFERENCES:
- See also: Related Info — http://www.kliniken-essen-mitte.de/leistung/fachabteilungen/naturheilkunde-u-integrative-medizin/home.html